CLINICAL TRIAL: NCT04850937
Title: Effect of Low-dose Esketamine on Postoperative Depression in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Ma Hong, Department of Anesthesiology, Yangzhou University Affiliated Hospital, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ES
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Depression
Keywords: Esketamine; Depression; pain; leptin
MeSH Terms: conditions — Depression; Pain | interventions — Esketamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: 180 patients will be divided into two groups according to the random number table method: control group (normal saline group),treatment group (esketamine group), 120 cases in each group.
Who Masked: Participant, Investigator
Masking Description: esketamine 10ml (5mg/ml) and normal saline 10ml were respectively set as drug A or drug B.
  Without the knowledge of the experimenter, the predetermined dose of drug A or B will be given to the experimenter before induction of anesthesia, with 0.05 mL /kg for each patient.
  After all samples are collected, the third party will announce the grouping and medication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Experimental): The experimental group will be given 0.25mg/kg esketamine slowly intravenously after anesthesia induction During administration, blood pressure and heart rate were observed.
  Interventions: Drug: Esketamine
- Group C (Placebo Comparator): The control group will receive the same amount of normal saline after anesthesia induction
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Esketamine — The experimental group will be given 0.25mg/kg esketamine slowly intravenously after anesthesia induction
  Arms: Group S
Drug: normal saline — The experimental group will be given 0.5ml/kg normal saline intravenously after anesthesia induction
  Arms: Group C

SUMMARY:
esketamine is an optical isomer of ketamine. Compared with ketamine, esketamine has the characteristics of higher effective value, stronger receptor affinity, less adverse reactions of nervous system, and pharmacokinetics is controllable.

Domestic and foreign studies have focused on the therapeutic effect of esketamine on major depression, but less attention has been paid to perioperative depression.This study intends to explore the effect of small doses of esketamine on patients with breast cancer.Postoperative depression and pain are observed.

DETAILED DESCRIPTION:
This study intends to explore the effect of small doses of esketamine on patients with breast cancer.WE pay attention to :

1. Safety of low-dose single intravenous injection of esketamine (1)The influence of intraoperative vital signs of patients after medication, such as blood pressure and heart rate fluctuation; (2)the duration of recovery after anesthesia; (3)postoperative adverse reactions, such as nausea and vomiting, dizziness and diplopia, respiratory depression, laryngeal spasm, delirium agitation, etc
2. Effect of single intravenous injection of low-dose ketamine on postoperative depression in patients undergoing radical mastectomy (1) 1 day before surgery, 2 days, 5 days, 30 days, 90 days after surgery Hamilton Depression Scale scores; (2) The serum leptin level 1 day before surgery, 2 days after surgery and 5 days after surgery; (3) Correlation between depression scale score and leptin level
3. Effects of low dose esketamine on acute and chronic pain in patients undergoing radical mastectomy

   * visual analogue scale scores at 6, 12 and 24 hours after surgery;

     * visual analogue scale scores at 3, 5, 30 and 90 days after surgery;

       * the number of analgesic remedies

ELIGIBILITY:
Inclusion Criteria:

* (1) Female patients who planned to undergo unilateral modified radical mastectomy in breast surgery; (2)Years of education ≥5 years,American Society of Anesthesiologists Ⅰ-II grade; (3) All patients undergoing surgery within 1 week after diagnosis of breast cancer, and do not receive preoperative radiotherapy or chemotherapy; (4) All the patients were married and had children, and were mainly cared for by their immediate family members after surgery.

Exclusion Criteria:

* (1) Antidepressant treatment was received within the last 2 months; (2) previous personality disorder, intellectual retardation, brain injury or brain disease, combined with schizophrenia, mania and other mental diseases; (3) Preoperative patients with hyperthyroidism or hypothyroidism, severe cardiovascular disease, diabetes, severe blood deficiency, and abnormal heart, lung, liver, and kidney functions; (4) with diseases of the immune system, or use drugs that have obvious effects on the immune system; (5) Pregnancy or lactation;

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 90 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
depression score | Change from Baseline score at 3 months
  The total rough score is the sum of all the scores in the 20 items, and then the rough score is multiplied by 1.25 to take the round part to get the standard score.
  An SDS score of 53 to 62 is classified as mild depression, 63 to 72 as moderate depression, and 73 or more as major depression.

SECONDARY OUTCOMES:
pain score | Change from Baseline score at 3 months
  visual analogue scale 0 points painless;
  1 to 3 points for mild pain; 4 to 6 points moderate pain; Severe pain on a 7-9 scale; 10 points severe pain.
The serum leptin level | Change from 1 day before surgery to 90 days after surgery
  The serum leptin level 1 day before surgery, 2 days ,5 days 30 days and 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: LIU M YU, Principal Investigator — Yangzhou University
Locations (1):
- Affiliated hospital of yangzhou university, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No